CLINICAL TRIAL: NCT03274713
Title: Efficacy of Electro-acupuncture Versus Manual Acupuncture for Knee Osteoarthritis: a Randomized Controlled Pilot Trial
Brief Title: Efficacy of Electro-acupuncture Versus Manual Acupuncture on Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: zhouping (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Jishuitan Hospital (Other)
Responsible Party: Sponsor-Investigator, zhouping, Postgraduate Student, Beijing Hospital of Traditional Chinese Medicine
Organization: Beijing Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017BL-020-01
Record Dates: First submitted 2017-08-30; First posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis Of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electro-acupuncture group (Experimental): After recruiting, patients are assigned to the electro-acupuncture group by randomization,and then receive electro-acupuncture treatment.Both treatments consist of 24 sessions of 30 minutes duration, administered over 8 weeks (usually three sessions per week). Participants in both groups will be evaluated at baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks.
  Interventions: Device: Electro-acupuncture
- Manual acupuncture group (Experimental): After recruiting, patients are assigned to the manual acupuncture group by randomization,and then receive manual acupuncture treatment.Both treatments consist of 24 sessions of 30 minutes duration, administered over 8 weeks (usually three sessions per week). Participants in both groups will be evaluated at baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks.
  Interventions: Device: Manual acupuncture

INTERVENTIONS:
Device: Electro-acupuncture — Patients in this group will be treated by use of 6-7 local acupuncture points (ST34, ST35, ST36, EX-LE2, EX-LE5, GB33, GB34, SP9, SP10, LR7, LR8 and Ashi) and 2-3 distal points (GB31, GB36, GB39, GB41, ST40, ST41, LR3, BL60, SP6 and KI3). Needles will be stimulated manually for 10 seconds to achieve "De Qi" sensation and an electrical apparatus (HANS-200A acupoint nerve stimulator, Nanjing Jisheng Medical Co., Ltd. production, wave of 2/100Hz) will be then connected to the needles with alligator clips to stimulate the needles in pairs ST36-SP9/GB34 and ST34-SP10. The stimulus intensity will be increased until the patient reports a strong but comfortable intensity.
  Arms: Electro-acupuncture group
Device: Manual acupuncture — Participants in the group have the same schedule as the electro-acupuncture group except that the electrical apparatus has working power indicator and sound without actual current output.
  Arms: Manual acupuncture group

SUMMARY:
Knee osteoarthritis (KOA), also called degenerative knee disease, is one of the most common bone and joint diseases in clinic. It often occurs in middle-aged people, especially women. It was estimated to affect more than 9 million individuals in the United States in 2005 and is a leading cause of disability and medical costs. Most elderly people over the age of 65 have radiographic and/or clinical evidence of osteoarthritis. KOA is a lifelong disease which can lead to obvious pain, joint stiffness, limitation of activity and even joint failure or disability.According to the papers published in the past years, we find that acupuncture therapy for the treatment of knee osteoarthritis include manual acupuncture, electro-acupuncture, acupotomy, laser acupuncture, fire needle and so on, among which manual acupuncture and electro-acupuncture are most commonly used.The aim of this study is to compare the effectiveness of electro-acupuncture and manual acupuncture in reducing pain and improving function in patients with KOA.

DETAILED DESCRIPTION:
Participants will be randomly allocated to one of two groups. Those in the first group receive electro-acupuncture, which involves having needles inserted into acupuncture points (locations on the body affected by acupuncture) which are stimulated manually for 10 seconds to create "De Qi" sensation and an electrical apparatus (HANS-200A acupoint nerve stimulator, Nanjing Jisheng Medical Co., Ltd. production, wave of 2/100Hz) was then connected to the needles with alligator clips to stimulate the needles in pairs ST36-SP9/GB34 and ST34-SP10. The stimulus intensity will be increased until the patient reported a strong but comfortable intensity. Those in the second group have the same schedule as the electro-acupuncture group except that the electrical apparatus has working power indicator and sound without actual current output. Both groups will receive 30-minute, 24 sessions intervention over eight weeks. Moreover, a number of questionnaires at the start of the study and then again after 4, 8, 12 and 16 week will be completed by participants.

It is expected that participants will benefit from a decrease in pain and improved function. The risks of participation are minimal. Occasionally, acupuncture can make people feel nauseous or experience a temporary increase in pain either during or after treatment. Rare side effects during acupuncture treatment include fainting, infection and subcutaneous hematoma (pooling of blood under the skin). Participants will be warned of these potential side-effects before consenting to have acupuncture.

Participants will be allowed, or required, to withdraw from the trial based on the following:

1. A major protocol violation;
2. Development of a serious disease preventing continuation in the trial;
3. Adverse events related to acupuncture;
4. Request to be withdrawn from the trial. The purpose is to accumulate clinical data, obtain the outcome data of the intervention method and prove the feasibility of the study protocol. Sixty patients will be selected as the sample size according to clinical experience.

ELIGIBILITY:
Inclusion Criteria:

* Age 45-75 years old, male or female
* Single / bilateral knee pain, duration of more than 6 months
* KL (Kellgren-Lawrence) grade Ⅱ or Ⅲ
* VAS ≥ 40mm
* Signed informed consent

Exclusion Criteria:

* Surgery history of knee or waiting for surgery (knee replacement or knee arthroscopy)
* History of arthroscopy within 1 year or intra-articular injection within 4 months
* Knee pain caused by other diseases (such as joint bodies, severe effusion of joint cavity, infection, malignant tumors, autoimmune diseases, trauma, etc.)
* Severe acute/chronic organic or mental diseases
* Coagulation disorders (such as hemophilia, etc.)
* Pregnant women, pregnant and lactating women
* History of receiving acupuncture or massage treatment within one month
* Participation in another clinical study in the past 3 months
* With a cardiac pacemaker, metal allergy or needle phobia

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
Success Rate | baseline, 8 weeks
  a change of 50% from baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) pain, stiffness and function scores at 8 weeks.

SECONDARY OUTCOMES:
Pain | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  using WOMAC pain subscale
Stiffness | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  using WOMAC stiffness subscale
Knee-joint function | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  using WOMAC functional subscale
Quality of life | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  using the 12-Item Short Form Health Survey (SF-12)
Number of emergency analgesics (Celebrex/Loxonin) used | baseline, 4 weeks, 8 weeks, 12 weeks and 16 weeks
  using Drug Use Form
Inflammatory markers | baseline, 8 weeks
  Luminex liquid chip method (LuminexxMAP, Technology, USA) Bio-plex200 system high throughput analysis platform (Bio-Rad) will be used to detect the expression of free protein in serum. Patients will receive fasting blood samples in the morning and then be centrifuged with 3000r/min, 15min in two hours.
Credibility/expectancy questionnaires | baseline
  Credibility/expectancy questionnaires are used to assess the credibility and expectancy of the patients
Adverse events | up to 16 weeks
  using Adverse Event Form

CONTACTS AND LOCATIONS:
Overall Officials: Cunzhi Liu, M.D, Study Director — Beijing Hospital of Traditional Chinese Medicine
Locations (1):
- Beijing Hostipal of Traditional Chinese Medicine affiliated to Capital medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shi GX, Tu JF, Wang TQ, Yang JW, Wang LQ, Lin LL, Wang Y, Li YT, Liu CZ. Effect of Electro-Acupuncture (EA) and Manual Acupuncture (MA) on Markers of Inflammation in Knee Osteoarthritis. J Pain Res. 2020 Aug 26;13:2171-2179. doi: 10.2147/JPR.S256950. eCollection 2020. PMID 32904642
- [Derived] Wang TQ, Li YT, Wang LQ, Shi GX, Tu JF, Yang JW, Hou YQ, Lin LL, Sun N, Zhao JJ, Hou HK, Liu CZ. Electroacupuncture versus manual acupuncture for knee osteoarthritis: a randomized controlled pilot trial. Acupunct Med. 2020 Oct;38(5):291-300. doi: 10.1177/0964528419900781. Epub 2020 Feb 5. PMID 32022581
- [Derived] Tu JF, Yang JW, Lin LL, Wang TQ, Du YZ, Liu ZS, Hu H, Zhao JJ, Yu XG, Jia CS, Wang J, Wang T, Hou YQ, Zou X, Wang Y, Shao JK, Wang LQ, Yu ZS, Liu CZ. Efficacy of electro-acupuncture and manual acupuncture versus sham acupuncture for knee osteoarthritis: study protocol for a randomised controlled trial. Trials. 2019 Jan 25;20(1):79. doi: 10.1186/s13063-018-3138-x. PMID 30683147